CLINICAL TRIAL: NCT01373307
Title: An Intergenerational CBPR Intervention to Reduce Appalachian Health Disparities
Brief Title: An Intergenerational Community Based Participatory Research (CBPR) Intervention to Reduce Appalachian Health Disparities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nancy Schoenberg (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Nancy Schoenberg, Sponsor/PI, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: R01DK081324 (NIH); R01DK081324 (NIH)
Record Dates: First submitted 2011-06-08; First posted 2011-06-14 (Estimated); Last update posted 2015-07-13 (Estimated); Status verified 2014-12

CONDITIONS: Overweight; Obesity
Keywords: Overweight; obesity; Appalachian; intergenerational; families; energy balance; group-randomized trial
MeSH Terms: conditions — Overweight; Obesity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early Intervention (Experimental): Participants are nested in churches which were randomly assigned to receive the intervention first.
  Interventions: Behavioral: LHA-delivered energy balance classes/activities
- Delayed Intervention (No Intervention): Wait-list control group. Participants are nested in churches which were randomly assigned to receive the intervention at a later date. Delayed Intervention participants receive an educational luncheon addressing stress reduction during the window of no intervention.

INTERVENTIONS:
Behavioral: LHA-delivered energy balance classes/activities — 4-6 sessions delivered by local LHA to age-appropriate groups (i.e., children/adolescents and adults), based on We Can! And Media Smart Youth curricula.
  Arms: Early Intervention

SUMMARY:
The study purpose is to evaluate the effectiveness of a culturally appropriate, faith-placed lay health advisor intervention aimed at increasing fruit and vegetable intake and physical activity among intergenerational Appalachian individuals and families.

DETAILED DESCRIPTION:
The developmental phase of this project incorporated community based participatory research (CBPR) principles to identify the needs and preferences of community members with regard to energy balance. In the intervention phase, this group-randomized trial administers and evaluates an intergenerational, culturally appropriate energy balance intervention aimed at increasing fruit and vegetable intake and increasing physical activity among participants in 6 distressed Appalachian counties. Faith institutions are recruited and randomized to treatment or wait-list control conditions, and participants are recruited and enrolled within those institutions. Focusing on Appalachian children, parents, and grandparents, local lay health advisors deliver a series of group presentations, adapted from We Can! and Media Smart Youth. In addition, the project provides culturally consonant leave-behind "booster" activities, including square dances, cooking classes, and community gardens.

ELIGIBILITY:
Inclusion Criteria:

* Age 8 years or above
* Able to provide informed consent/assent

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1250 (Actual)
Dates: Start 2010-03; Primary Completion 2012-07 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change in self-reported fruit and vegetable intake from baseline | Assessed approximately 4 months after baseline
  Amount of fruit and vegetable intake is measured using an FFQ, pretested in focus groups comprised of members of the target population. Positive change (i.e., increasing fruit and vegetable intake) from baseline to post-test will be coded as "1," while negative or no change will be coded "0." This assessment occurs after the Early Treatment group has completed the intervention.
Change in self-reported physical activity from baseline | Assessed at approximately 4 months after baseline
  Amount of physical activity is measured using instruments with demonstrated reliability and validity, pretested in focus groups comprised of members of the target population. Positive change (i.e., increasing physical activity) from baseline to post-test will be coded as "1," while negative or no change will be coded "0." This assessment occurs after the Early Treatment group has completed the intervention.
Change in body mass index (BMI) from baseline | Assessed at approximately 4 months after baseline
  Positive change (i.e., decreasing BMI when indicated, or maintaining BMI when not indicated) from baseline to post-test will be coded as "1," while negative or no change will be coded "0." This assessment occurs after the Early Treatment group has completed the intervention.

SECONDARY OUTCOMES:
Change in stage of readiness to change each health behavior (i.e., fruit and vegetable intake, physical activity) from baseline | Assessed approximately 4 months after baseline
  Stage of readiness to change is measured using instruments with demonstrated reliability and validity, pretested in focus groups comprised of members of the target population. Positive change in stage of readiness from baseline to post-test will be coded as "1," while negative or no change will be coded "0." This assessment occurs after the Early Treatment group has completed the intervention.
Number of visits completed | Approximately 4 months after baseline
  This process measure will reflect the number of visits/classes attended by participants, as a means of assessing participation rate and feasibility.
Retention (i.e., number of participants who complete all planned assessment timepoints) | Approximately one year after baseline
  Retention numbers will be assessed as a process measure outcome. Participants who complete all study assessment timepoints will be coded as "1," while participants who drop out will be coded "0." Number/percentage of participants who remained enrolled and complete all study procedures and assessments will be used as an indicator of feasibility in the community setting.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Schoenberg, Ph.D., Principal Investigator — University of Kentucky
Locations (1):
- Faith Moves Mountains, Whitesburg, Kentucky, United States